CLINICAL TRIAL: NCT04326140
Title: Robot-assisted Therapy Combined With Mirror Priming in Upper Limb Training in Stroke: Randomized Clinical Trial and Neuromuscular Mechanism
Brief Title: Robot-assisted Therapy Combined With Mirror Priming in Upper Limb Training in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201801525B0
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Stroke
Keywords: Robot assisted therapy; mirror priming; upper limb; neuromuscular mechanism
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic training with mirror therapy (Experimental): Participants will receive 18 intervention sessions for about 6 consecutive weeks in a clinical setting (1 hour per session, 3 sessions per week). For each intervention session, participants will first receive 20 minutes mirror therapy followed by 40 minutes robotic-assisted training (robotic-assisted training includes 10 minutes active/passive training mode and 30 minutes robot-participant interactive training mode).
  Interventions: Device: mirror therapy; Device: robotic-assisted training
- Robotic-assisted training (Sham Comparator): The training procedure will be the same as the robotic-assisted training with mirror therapy group except that sham mirror therapy will be provided in the first 20 minutes in the intervention session.
  Interventions: Device: robotic-assisted training; Device: sham mirror therapy

INTERVENTIONS:
Device: mirror therapy — The affected side wears the machine, assists by the machine, and performs the same action with the good hand. According to the posture condition, selects two suitable actions in the three actions (all fingers open, all fingers close, all fingers open and close). The action is 10 minutes each.
  Arms: Robotic training with mirror therapy
Device: robotic-assisted training — The hand brace is worn on the dorsal side of the impaired hand with 2 surface sensors attached to the extensor and flexor muscles of the arm to detect the surface electromyographic signals (sEMG) for active participation during exercise. The sEMG signals are processed so the patient can visualise the active movement of the muscle where sEMG electrodes are positioned. Different training modes allow the therapist to customise the level of assistance that the Hand of Hope provides. The difficulty level of each mode can be adjusted according to the patient's need.
Device: sham mirror therapy — The mirror was masked. The intervention was the same as the mirror therapy.
  Arms: Robotic-assisted training

SUMMARY:
This project will employ the robot-assisted system to assist patients to perform the grasping and releasing movement of both hands simultaneously while mirror priming strategy is applied, and, then, perform intensive and game-based finger movement training with the robotic assistance. This randomized controlled trial is the first study to explore the benefits of combined robotic-assisted therapy and mirror priming strategy in stroke patients. This proposed combined approach might be a novel combination of enhancing movement performance, daily function and quality of life for patients with stroke.

DETAILED DESCRIPTION:
Approximately 70% to 80 % of stroke patients suffered from upper limb (UE) hemiparesis which limited their daily function and quality of life, as well as required considerable demands of long-term medical care. Robot-assisted training and mirror priming has been advocated as part of contemporary approaches. The robotic-assisted therapy mainly emphasized on the proximal part of UE, such as shoulder and elbow movement. While mirror priming strategy has been increasingly employed in the UE training, one question has been raised: the affected UE of stroke patients cannot complete the same movement as the sounded limb synchronously. This project will employ the robot-assisted system to assist patients to perform the grasping and releasing movement of both hands simultaneously while mirror priming strategy is applied, and, then, perform intensive and game-based finger movement training with the robotic assistance. This randomized controlled trial is the first study to explore the benefits of combined robotic-assisted therapy and mirror priming strategy in stroke patients. This proposed combined approach might be a novel combination of enhancing movement performance, daily function and quality of life for patients with stroke. This project will further explore the possible neuro-muscular mechanism underlying this combined mirror priming with robotic training. This project attempts to compare the cortical activation and neuromuscular control of patients with stroke and age-matched healthy adults in terms of electroencephalography (EEG) and muscle tone measurement. The findings of this study may lay an evidence-based foundation for bridging basic science and clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Stroke more than 3 months.
* Modified Ashworth Scale proximal part ≤ 3, Modified Ashworth Scale distal part ≤ 2, and no serious muscle spasms.
* The myoelectric signal can be detected to activate the instrument
* Unilateral paresis (FMA score<60)
* No serious cognitive impairment (i.e., Mini Mental State Exam score > 24)
* Can provide informed consent

Exclusion Criteria:

* Other neurological disease
* Complete sense of body defect
* Inability to understand instructions
* current participation in any other research
* Botulinum Toxin injection within 3 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change scores of Fugl-Myer Assessment (FMA) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The upper-extremity subscale of the FMA will be used to assess motor impairment. There are 33 upper extremity items measuring the movements and reflexes of the shoulder/elbow/forearm, wrist, hand, and coordination/speed. Each score is on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully). The maximum score is 66, indicating optimal recovery. The subscore of a proximal shoulder/elbow (FMA s/e: 0-42) and a distal hand/wrist (FMA h/w: 0-24) will be calculated to investigate the treatment effects on separate upper extremity elements. The FMA has good reliability, validity, and responsiveness in stroke patients.
Change scores of Active Range of Motion (AROM) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  Patient performs the exercise to move the joint without any assistance to the muscles surrounding the joint.
Change scores of grip and pinch power | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Jamar hand dynamometer is the most widely cited in the literature and accepted as the gold standard by which other dynamometers are evaluated. Excellent concurrent validity of the Jamar hand dynamometer is reported. The Jamar hand dynamometer measure the grip-strength. The norm of healthy male aged 18 to 75 years is from 64.8 lb to 121.8 lb, while the norm of healthy female aged 18 to 75 years is from 41.5 lb to 78.7 lb. Higher value represent a greater grip-strength.
Change scores of Modified Ashworth Scale (MAS) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The MAS is a 6-point ordinal scale that measures muscle spasticity in patients with brain lesions. Higher score indicates higher muscle tone. Investigators will assess the MAS scores of UE muscles, including biceps, triceps, wrist flexors and extensors, and finger flexors and extensors. The validity and reliability of MAS for patients with stroke were established to be adequate to good.
Change scores of Medical Research Council scale (MRC) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The MRC is an ordinal scale that assesses muscle strength. The scoring for each muscle ranges from 0 to 5, with a higher score indicates stronger muscle. The reliability of MRC for all muscle groups was good to excellent in patients with stroke.
Change scores of Revised Nottingham Sensory Assessment (rNSA) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The rNSA includes tactile sensation, kinesthetic sensation, and stereognosis. The rNSA is reliable measure of sensory function in stroke patients. For tactile sensation, the patient will be asked to indicate whenever he or she feels the test sensation. For kinesthetic sensations, all 3 aspects of movement will be tested: appreciation of movement, its direction and accurate joint position sense. The limb on the affected side of the body will be supported and moved by the examiner in various directions but movement is only at one joint at a time. The patients will be asked to mirror the change of movement with the other limb. For stereognosis, the object will be placed in the patient's hand for a maximum of 30 seconds. Identification is by naming, description or by pair-matching with an identical set. The object may be moved around the affected hand by the examiner. The rNSA has good intrarater and interrater reliability (Lincoln, Jackson, & Adams, 1998).
Change scores of Wolf Motor Function Test (WMFT) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The WMFT was designed to assess the effects of CIT on arm function after stroke and traumatic brain injury (Wolf, Lecraw, Barton, & Jann, 1989). There are 15 function-based and 2 strength-based tasks. For timed functional tasks, completion times from 0 to 120 seconds are averaged. For functional ability scoring, 6-point ordinal scales are used, where 0 indicates "does not attempt with the involved arm" and 5 indicates "arm does participate, movement appears to be normal." The clinimetrics of the WMFT has been ascertained in stroke patients.
Change scores of 10-Meter Walk Test (10MWT) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  We include this test because improvement in UL motor control may contribute to arm swing and help generate forward propulsion at the foot (Tester, Barbeau, Howland, Cantrell, & Behrman, 2012) and may improve mobility and functional ambulation (Lin, et al., 2009). The 10MWT assess mobility function by measuring the time and the numbers of strides required to walk 10 meters under two conditions: (1) with the self-pace of each participant (self-pace); (2) with the speed that the participants walked as soon as possible (Rossier & Wade, 2001). The velocity and stride length of the participant are calculated. Research has validated the 10MWT in measuring mobility in stroke.
Electromyography (EMG) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  Raw EMG activities from the muscles of interest during unilateral and bilateral reaching while the patient is sitting and standing will be recorded using the AcqKnowledge data analysis software.
Change scores of Mini-Mental State Exam (MMSE) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Mini-Mental State Examination (MMSE) is the most commonly administered psychometric screening assessment of cognitive functioning. The MMSE is used to screen patients for cognitive impairment, track changes in cognitive functioning over time, and often to assess the effects of therapeutic agents on cognitive function. The total score of MMSE ranged from 0 to 30. Higher values represent a better cognitive functioning.
Change scores of Montreal Cognitive Assessment (MoCA) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Montreal Cognitive Assessment (MoCA) will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitvie functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Motor Activity Log (MAL) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The MAL consists of 30 structured questions to interview how the patients rate the frequency (amount of use subscale) and quality (quality of movement subscale) of movements while using their affected arm to accomplish each of the 30 daily activities. The score of each item ranges from 0 to 5, and the higher scores indicate more frequently used or higher quality of movements. The clinimetric properties of the MAL in stroke patients have been validated (Uswatte, Taub, Morris, Light, & Thompson, 2006).
Change scores of Nottingham Extended Activities of Daily Living Scale (NEADL) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The NEADL scale is a measure of Instrumental ADL ability, comprising sub-scales for mobility, household ability and leisure activity. The NEADL consists of 22 activity items, scoring on the basis of the required level of assistance. The range of total score is 0-66, and higher score representing better function. This measure is administered 3 times during the study period.
Change scores of Stroke Impact Scale (SIS) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The SIS 3.0 is a stroke-specific instrument of health-related quality of life. It contains 59 items measuring 8 domains (i.e., strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion. memory and thinking and participation) with a single item assessing perceived overall recovery from stroke. Items are rated on a 5-point Likert scale with lower scores indicating greater difficulty in task completion during the past week. The reliability, validity, and responsiveness have been shown to be satisfactory in stroke patients.
Change scores of stroke self-efficacy questionnaire (SSEQ) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  the Stroke Self-Efficacy Questionnaire (SSEQ) , a questionnaire developed to measure the most relevant self-efficacy and self-management domains specific to the stroke population. It contains 13 items that are rated on a 0 - 10 scale, with higher scores indicating greater levels of self-efficacy. Questionnaire includes a range of relevant functional tasks such as walking, getting comfortable in bed, as well as some self-management tasks.
Change scores of Daily Living Self-Efficacy Scale (DLSES) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The DLSES is designed to measure self-efficacy in psychosocial functioning and self-efficacy in activities of daily living, regardless of level of physical impairment.
Change scores of Functional Abilities Confidence Scale (FACS) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Functional Abilities Confidence Scale (FACS) was designed to measure the degree of self-efficacy or confidence a patient exhibits with various movements or postures.
Kinematic analysis | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The kinematic analysis will involve unilateral and bilateral tasks, in which the participants will be asked to perform by using the affected upper limb or both upper limb simultaneously. A motion analysis system with 7 cameras (VICON MX 30d, Oxford Metrics Inc., Oxford, UK) will be used to capture the motion of arm (s) in kinematic testing. The markers will be attached on the styloid processes of the ulna. Depending on the unilateral or bilateral tasks, the makers will be placed on the affected arm or the both arms, respectively.
Task-based Electroencephalogram (EEG) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Task-based EEG will be collected when participants perform the n-back task before and after the intervention program to examine the effects of training on neural plasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan